CLINICAL TRIAL: NCT06006975
Title: R&D of Innovative Technology for Predicting and Early Warning of Delayed Cerebral Ischemia After Subarachnoid Hemorrhage
Brief Title: Early Warning of Delayed Cerebral Ischemia
Acronym: EWoDCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Collaborators: Kaunas University of Technology (Other); Lithuanian University of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: EWoDCI ver.C; 01.2.2-LMT-K-718-03-0091 (Other Grant/Funding Number: Research Council of Lithuania)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Vasospasm, Cerebral; Ischemia; Outcome, Fatal
Keywords: subarachnoid hemorrhage; delayed cerebral ischemia; computed tomography
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subarachnoid hemorrhage (SAH) patients: Patients after aneurysmal subarachnoid hemorrhage who received routine treatment (aneurysm clipping surgery, post operative care and multimodal monitoring in ICU).
  Interventions: Radiation: Computed Tomography (CT) and Computed Tomography Angiography (CTA); Diagnostic Test: Multimodal physiological monitoring

INTERVENTIONS:
Radiation: Computed Tomography (CT) and Computed Tomography Angiography (CTA) — CT and CTA examinations are performed as a routine procedure to evaluate SAH severity and to diagnose cerebral vasospams and delayed cerebral ischemia.
Diagnostic Test: Multimodal physiological monitoring — Patients are monitored routinely during their treatment in ICU. Multimodal physiological monitoring include continuous monitoring of arterial blood pressure (ABP), intracranial pressure (ICP) (if available), ETCO2 (if available), cerebral perfusion pressure (if available), cerebral blood flow velocity (CBFV) measured in middle cerebral artery and heart rate.
  Non invasive CBFV will be measured by using TCD device DWL Multi Dop-T. Invasive ICP will be measured by using Codman ICP Express or Raumedic ICP monitor.

SUMMARY:
The goal of this observational study is to learn about the possibility to predict clinical course of subarachnoid hemorrhage (SAH) patients by performing the retrospective analysis of clinical data available in early pre-vasospasm phase.

The main questions it aims to answer are:

* What biomarkers retrieved from Computed Tomography (CT) and Computed Tomography Angiography (SAH location, leaked blood volume, cerebrospinal fluid volume, etc.) can be used to predict development of cerebral vasospasms, delayed cerebral ischemia and patients' outcome.
* What biomarkers retrieved from transcranial Doppler examinations in early pre vasospasm can be used to predict development of cerebral vasospasms, delayed cerebral ischemia and patients' outcome.
* What biomarkers retrieved from multimodal physiological monitoring in early pre vasospasm can be used to predict development of cerebral vasospasms, delayed cerebral ischemia and patients' outcome.
* What is impact of other clinical data (blood test results, age, gender, etc.) on development of cerebral vasospasms and delayed cerebral ischemia.

DETAILED DESCRIPTION:
An adequate timely prognosis of cerebral vasospasms and delayed cerebral ischemia (DCI) occuring after spontaneous aneurysmal subarachnoid haemorrhage (aSAH), is vitally essential to selecting an individualized and timely treatment strategy. Cerebral vasospasms (CV) occur in up to 70% of aSAH cases, and in two thirds of those cases DCI develops, thus increasing the mortality rate up to 50%. Every year up to 770 000 people suffer from aSAH and receive neurosurgical treatment. Because of a large amount of factors (blood leak volume and its distribution in the subarachnoid space, reactivity of cerebral blood vessels, biochemical blood composition and demographical factors) and their complex interactions to contribute the development of CV/DCI, currently there are no reliable methods and technologies allowing reliably prediction of the consequences of SAH.

For a more effective treatment of aSAH patients an innovative method for early warning of CV and DCI phenomena is offered. The method is based on identifying of the associations of different physiological modalities and prognostic factors with the SAH patients' outcome (factors the obtained from CT images analysis, numerical modelling of SAH evolution and multimodal cerebral hemodynamics monitoring).

The goal of this observational study is to learn about the possibility to predict clinical course of subarachnoid hemorrhage (SAH) patients by performing the retrospective analysis of clinical data available in early pre-vasospasm phase.

The main questions it aims to answer are:

* What biomarkers retrieved from Computed Tomography (CT) and Computed Tomography Angiography (SAH location, leaked blood volume, cerebrospinal fluid volume, etc.) can be used to predict development of cerebral vasospasms, delayed cerebral ischemia and patients' outcome.
* What biomarkers retrieved from transcranial Doppler examinations in early pre-vasospasm can be used to predict development of cerebral vasospasms, delayed cerebral ischemia and patients' outcome.
* What biomarkers retrieved from multimodal physiological monitoring in early pre vasospasm can be used to predict development of cerebral vasospasms, delayed cerebral ischemia and patients' outcome.
* What is impact of other clinical data (blood test results, age, gender, etc.) into development of cerebral vasospasms, delayed cerebral ischemia.

Study objectives:

1. To perform retrospective analysis neuroradiological examination data (CT/CTA images) of patients who experienced spontaneous aSAH, by identifying factors that allow early prediction of CV and DCI
2. To perform retrospective analysis of the collected data of multimodal brain physiological monitoring (intracranial pressure, arterial blood pressure, cerebral blood flow velocity, heart rate) by determining the factors that allow to predict CV and DCI.
3. To perform retrospective analysis of other clinical data (blood test results), demographic data (gender, age) and their impact on development of CV and DCI.
4. To develop the algorithm of predicting of CV, DCI and patients' outcome based on the accumulated neuroradiological examination and multimodal monitoring data.

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid hemorrhage patients who require SAH surgery and post-operative routine treatment.

Exclusion Criteria:

* persons with mental disorders, but who can give consent to participate in biomedical research;
* minors;
* students, if their participation in biomedical research is related to studies;
* persons living in care institutions;
* soldiers during their actual military service;
* employees of health care institutions where biomedical research is conducted, subordinate to the researcher;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients treated at Vilnius University Hospital Santaros Klinikos that undergo brain surgery after subarachnoid hemorrhage (SAH) and routine post-operative treatment in ICU.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Cerebral vasospasms | CTA is performed routinely on 7th day after SAH or within period of 3-21 day after SAH if necessary
  Cerebral vasospasms are diagnosed by performing Computed Tomography Angiography (CTA) according to reduced diameters of cerebral arteries.
Delayed cerebral ischemia | CT is performed routinely on 7th day after SAH or within period of 3-21 day after SAH if necessary
  Delayed cerebral ischemia is diagnosed by performing Computed Tomography (CT)
Patient outcome | GOS is evaluated at discharge from hospital and after 30 days after SAH
  Patients' outcome is evaluated according to Glasgow Outcome Score (GOS). GOS scores are: 1 - death, 2 - persistent vegetative state, 3 - severe disability, 4 - moderate disability, 5 - low disability

CONTACTS AND LOCATIONS:
Overall Officials: Saulius Rocka, Prof. Dr., Principal Investigator — Clinic of Neurology and Neurosurgery, Faculty of Medicine, Vilnius University
Locations (1):
- Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No